CLINICAL TRIAL: NCT01304472
Title: Prasugrel Versus High Dose Clopidogrel in Patients With Stable Coronary Artery Disease and High Platelet Reactivity While on Chronic Clopidogrel Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-3
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: coronary angioplasty; clopidogrel resistance; prasugrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental): Prasugrel 10mg per day
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10mg per day
  Arms: Prasugrel
Drug: Clopidogrel — Clopidogrel 150mg per day
  Arms: Clopidogrel

SUMMARY:
Clopidogrel administration is considered standard of care in patients with stable coronary artery disease post PCI. However , a significant proportion of patients is considered clopidogrel resistant and this is shown to be accompanied by future adverse events. The hypothesis of the study is to define among consecutive outpatient clinics individuals with stable coronary artery disease being on chronic clopidogrel treatment, those that are clopidogrel resistant, as assessed with the VerifyNow point of care assay. Clopidogrel resistant patients will be randomized in a 1:1 fashion to either prasugrel 10mg or clopidogrel 150mg daily. Platelet reactivity will be assessed at Day 14, when treatment crossover will be performed without a washout period. At Day 28 platelet reactivity will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patients with history of coronary artery disease under chronic (≥ 6 months) clopidogrel treatment
* High on-clopidogrel platelet reactivity (≥235 Platelet Reactivity Units as assessed with the VerifyNow assay)
* Written Informed Consent

Exclusion Criteria:

* History of bleeding diathesis
* History of active bleeding within 6 months before randomization
* Chronic oral anticoagulation treatment
* Contraindications to antiplatelet treatment
* Known platelet function disorders
* Acute coronary syndrome within 30 days before randomization
* Cardiogenic shock
* Planned Percutaneous Coronary Intervention in the next 30 days
* Cancer
* Haemodialysis
* Platelet count < 100000/μL
* Hematocrit < 30%
* High likelihood of being unavailable on the Day 28 visit
* History of stroke
* Known allergy to clopidogrel and/or prasugrel

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in Platelet Reactivity | At 14 and 28 days after randomization
  Platelet reactivity in Platelet Reactivity Units (PRU) as assessed with the VerifyNow point of care assay will be measured at the end of the two treatment periods, namely at 14 and 28 days after randomization

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Dimitrios Alexopoulos, Pátrai
  - Patras University Hospital Cardiology Department, Pátrai